CLINICAL TRIAL: NCT02361463
Title: 2D Versus 3D Laparoscopic Training on a Virtual Reality Simulator - A Randomised Trial
Brief Title: 2D Versus 3D Laparoscopic Training on a Virtual Reality Simulator
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Stine Maya Dreier Sørensen, Master student / B.M.Sc., Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2015-001
Record Dates: First submitted 2015-02-03; First posted 2015-02-11 (Estimated); Last update posted 2018-10-02 (Actual); Status verified 2018-10

CONDITIONS: Stereoscopic Vision
Keywords: Laparoscopy;; Training;; Three-Dimensional

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 3D group (Experimental): Will practice under 3D vision conditions on a laparoscopic virtual reality simulator
  Interventions: Device: 3D vision
- 2D group (Active Comparator): Will practice under 2D vision conditions on a laparoscopic virtual reality simulator
  Interventions: Device: 2D vision

INTERVENTIONS:
Device: 3D vision — Laparoscopic simulator training to proficiency under 3D conditions
  Arms: 3D group
Device: 2D vision — Laparoscopic simulator training to proficiency under 2D conditions
  Arms: 2D group

SUMMARY:
Laparoscopy training programs with virtual reality simulators are widely used before new surgeons are allowed to operate on patients. Laparoscopic surgery results in shorter time to recover, less surgical trauma and thereby a shorter stay at the hospital compared with open surgery. However, it is more difficult to learn laparoscopic surgery, than open surgery, in part because surgeons have to work in a 3-dimensional space, through a 2-dimensional interface on a screen. This results in loss of depth perception and therefore a higher visual and cognitive load. This trial examines if using 3D vision instead of 2D vision on the laparoscopic virtual reality simulator reduces the time to reach proficiency, by decreasing the cognitive and visual load during practice on a Virtual Reality Simulator.

ELIGIBILITY:
Inclusion Criteria:

* Residents working in Denmark. Participants are required to have a medical license and provide informed consent before inclusion

Exclusion Criteria:

1. Participation in prior studies involving laparoscopic training.
2. Experience with laparoscopy surgery (having performed minimum one laparoscopic procedure as primary surgeon, including supervised procedures).
3. Performing more than 3 supervised laparoscopy surgeries during the intervention.
4. Performing laparoscopy surgery between the intervention and the retention test 3-6 weeks after.
5. No informed consent.
6. Does not speak Danish on a conversational level.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2015-02; Primary Completion 2015-06 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Time (minutes) to reach the predefined proficiency level for the basic skills and the salpingectomy procedure | 1 year

SECONDARY OUTCOMES:
Time (minutes) to reach the predefined proficiency level for the basic skills and salpingectomy procedure under 2D conditions after 3-6 weeks without laparoscopic training during the follow-up period | 1 year

OTHER OUTCOMES:
Workload: NASA TLX questionnaire after the first and fifth attempt on procedural module, | 1 year
Visual and physical discomfort questionnaire after each training session (adverse effect: eye strain, headache, dizziness, nausea, tired and sore neck/back), | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Stine Maya Dreier Sørensen, B.M.Sc., Principal Investigator — Centre for Clinical Education
Locations (1):
- Centre for Clinical Education, Copenhagen, Denmark

REFERENCES:
- [Background] Lusch A, Bucur PL, Menhadji AD, Okhunov Z, Liss MA, Perez-Lanzac A, McDougall EM, Landman J. Evaluation of the impact of three-dimensional vision on laparoscopic performance. J Endourol. 2014 Feb;28(2):261-6. doi: 10.1089/end.2013.0344. Epub 2014 Jan 10. PMID 24059674
- [Background] Votanopoulos K, Brunicardi FC, Thornby J, Bellows CF. Impact of three-dimensional vision in laparoscopic training. World J Surg. 2008 Jan;32(1):110-8. doi: 10.1007/s00268-007-9253-6. PMID 17992561
- [Background] Smith R, Schwab K, Day A, Rockall T, Ballard K, Bailey M, Jourdan I. Effect of passive polarizing three-dimensional displays on surgical performance for experienced laparoscopic surgeons. Br J Surg. 2014 Oct;101(11):1453-9. doi: 10.1002/bjs.9601. Epub 2014 Aug 18. PMID 25131843
- [Background] Alaraimi B, El Bakbak W, Sarker S, Makkiyah S, Al-Marzouq A, Goriparthi R, Bouhelal A, Quan V, Patel B. A randomized prospective study comparing acquisition of laparoscopic skills in three-dimensional (3D) vs. two-dimensional (2D) laparoscopy. World J Surg. 2014 Nov;38(11):2746-52. doi: 10.1007/s00268-014-2674-0. PMID 25002241
- [Background] Wilhelm D, Reiser S, Kohn N, Witte M, Leiner U, Muhlbach L, Ruschin D, Reiner W, Feussner H. Comparative evaluation of HD 2D/3D laparoscopic monitors and benchmarking to a theoretically ideal 3D pseudodisplay: even well-experienced laparoscopists perform better with 3D. Surg Endosc. 2014 Aug;28(8):2387-97. doi: 10.1007/s00464-014-3487-9. Epub 2014 Mar 21. PMID 24651895
- [Background] Cicione A, Autorino R, Breda A, De Sio M, Damiano R, Fusco F, Greco F, Carvalho-Dias E, Mota P, Nogueira C, Pinho P, Mirone V, Correia-Pinto J, Rassweiler J, Lima E. Three-dimensional vs standard laparoscopy: comparative assessment using a validated program for laparoscopic urologic skills. Urology. 2013 Dec;82(6):1444-50. doi: 10.1016/j.urology.2013.07.047. Epub 2013 Oct 2. PMID 24094658
- [Background] Mistry M, Roach VA, Wilson TD. Application of stereoscopic visualization on surgical skill acquisition in novices. J Surg Educ. 2013 Sep-Oct;70(5):563-70. doi: 10.1016/j.jsurg.2013.04.006. Epub 2013 May 20. PMID 24016365
- [Derived] Sorensen SMD, Konge L, Bjerrum F. 3D vision accelerates laparoscopic proficiency and skills are transferable to 2D conditions: A randomized trial. Am J Surg. 2017 Jul;214(1):63-68. doi: 10.1016/j.amjsurg.2017.03.001. Epub 2017 Mar 9. PMID 28302275